CLINICAL TRIAL: NCT02770092
Title: Anabolic Responsiveness to Protein Intake in Chronic Heart Failure and Chronic Obstructive Pulmonary Disorder
Brief Title: CHF COPD Sip Feed Anabolic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB2015-0676
Record Dates: First submitted 2016-05-05; First posted 2016-05-12 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Congestive Heart Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy (Experimental): screening visit: body weight and composition by DXA, height, and vital signs will be assessed.
  study day(s): may include combinations of stable isotope infusions and sip feeding with blood draws and cognition testing
  Interventions: Other: sip feeding with stable isotope infusion
- Chronic Obstructive Pulmonary Disorder (Experimental): screening visit: body weight and composition by DXA, height, and vital signs will be assessed.
  study day(s): may include combinations of stable isotope infusions and sip feeding with blood draws and cognition testing
  Interventions: Other: sip feeding with stable isotope infusion
- Congestive Heart Failure (Experimental): screening visit: body weight and composition by DXA, height, and vital signs will be assessed.
  study day(s): may include combinations of stable isotope infusions and sip feeding with blood draws and cognition testing
  Interventions: Other: sip feeding with stable isotope infusion

INTERVENTIONS:
Other: sip feeding with stable isotope infusion — such as glycerol, D2O, tyrosine, phenylalanine, glucose, arginine, and citrulline

SUMMARY:
Weight loss commonly occurs in patients with chronic heart failure (CHF) and chronic obstructive pulmonary disorder (COPD), negatively influencing their quality of life, treatment response and survival. Loss of muscle protein is generally a central component of weight loss in CHF and COPD patients, but patients also have reductions in fat mass and bone density, independent of the severity of the disease state. The purpose of this study is to provide detailed insight in disease related gut function by obtaining information on gut permeability, digestion and absorption of glucose, fat and protein in CHF and COPD patients compared to matched healthy controls. This will provide required information that is necessary to implement new strategies to develop optimal nutritional regimen in CHF and COPD.

DETAILED DESCRIPTION:
General aims:

* To study the whole-body protein anabolic effect of several dosages of a high-quality protein sip feeding in COPD and CHF subjects as compared to healthy controls.
* To investigate the anabolic threshold in subjects with COPD and CHF as compared to healthy controls.

Purpose and objectives: Although the Researchers' previous study supports the concept of supplementing high-quality milk proteins in chronic wasting diseases i.e., COPD and CHF, the dose-response anabolic effects of proteins with high EAA levels are still unclear. Furthermore, there is no insight in the actual protein requirements in COPD and CHF. The knowledge gained from this study will benefit insight in terms of promotion of protein gain after feeding in COPD and CHF subjects. Based on the obtained data of protein behavior (protein kinetics) the Researchers will be able to further refine and personalize nutritional supplementation in COPD and CHF subjects in order to stop and even restore progressive muscle wasting.

ELIGIBILITY:
Inclusion criteria CHF subjects:

* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lie in supine or elevated position for 8 hours
* Diagnosis of CHF; under regular care by cardiologist
* Reduced ejection fraction (<45%) assessed in the past 2 years
* NYHA class II-IV
* Clinically stable condition; no hospitalization 4 weeks preceding first study day
* Willingness and ability to comply with the protocol

Inclusion criteria COPD subjects:

* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lie in supine or elevated position for 8 hours
* Diagnosis of moderate to very severe chronic airflow limitation and compliant to the following criteria: FEV1 < 70% of reference FEV1
* Clinically stable condition and not suffering from a respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding year) at least 4 weeks prior to the first test day
* Shortness of breath on exertion
* Willingness and ability to comply with the protocol

Inclusion criteria healthy subjects:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Age 45 years or older (older control group)
* Age between 20-30 years old (young group)
* Ability to lay in supine or elevated position for 8 hours
* No diagnosis of CHF or COPD
* Willingness and ability to comply with the protocol

Exclusion Criteria all subjects:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (healthy subjects only)
* Established diagnosis of malignancy
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Body mass index >40 kg/m2 (healthy subjects only)
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* Use of protein or amino acid containing nutritional supplements within 5 days of first study day
* Current Use of long-term oral corticosteroids (CHF only)
* Use of short course of oral corticosteroids within 4 weeks preceding first study day
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* (Possible) pregnancy
* Already enrolled in another clinical trial and that clinical trial interferes with participating in this study

When during the period from enrollment to the test day any condition causing the subject to not meet inclusion criteria or to meet exclusion criteria, the subject will be excluded from the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Change in net whole-body protein synthesis | 0, 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210, 225, 240, 260, 280, 300, 320, 340, 360 ± 5 min
  Change in whole-body protein synthesis rate after intake of meal

SECONDARY OUTCOMES:
Body Composition | 15 minutes on screening or study day 1
  Body composition as measured by Dual-Energy X-ray Absorptiometry
Skeletal muscle strength | on study day 1
  handgrip and kin-com 1-leg test
Respiratory muscle strength | on study day 1
  Maximum inhalation and exhalation pressure
Gut function | In postabsorptive and prandial state every 20 minutes up to 6 hours before each sip feeding on study day
  Digestion of the stable tracers of amino acid
Group differences in state of mood as measured by the Hospital Anxiety and Depression Scale (HADS) | Postabsorptive state during 3 hours and change after feeding on study day 1
  a fourteen item self-assessment scale. Seven of the items related to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression.
Executive Function-Adolescent/Adult Sensory Profile (ASP): | Postabsorptive state during 3 hours and change after feeding on study day 1
  a standardized self-questionnaire that generates an individualized profile of sensory processing across four quadrants: low registration, sensation seeking, sensory sensitivity, and sensation avoiding.
Group differences in quality of life as measured by Short Form (36) Health Survey (SF36) | Postabsorptive state during 3 hours and change after feeding on study day 1
  self administered questionnaire that measures each of the following eight health concepts: Physical Functioning (PF); Role-Physical (RP); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Role-Emotional (RE); Mental Health (MH) as well as a reported Health Transition item (HT).
Group differences in activity as measured by Physical Activity Scale for the Elderly (PASE) | Postabsorptive state during 3 hours and change after feeding on study day 1
  questionnaire is intended for use in an elderly population and focuses on 3 types of activities: leisure time activities, household activities and work-related activities.
Group differences in attention and executive functions as measured by Stroop Color-Word Test (SCWT), | Postabsorptive state during 3 hours and change after feeding on study day 1
  a word page with words printed in black ink, a color page with blocks printed in color, and a color-word page where the color and the word do not match. The examinee reads the words or names the ink colors as quickly as possible within a time limit. Measures selective attention and inhibitory control. The total time in seconds was reported for each trial.
Group differences in state of mood as measured by the Profile of Mood State (POMS) | Postabsorptive state during 3 hours and change after feeding on study day 1
  A psychological distress scale to measure mood disturbance in 6 domains - fatigue-inertia, vigor-activity, tension-anxiety, depression-dejection, anger-hostility, and confusion-bewilderment. Healthy populations take 3 to 7 minutes to complete, and others may take up a bit longer.
Group differences in learning and memory as measured by Controlled Oral Word Association Test (COWAT), | Postabsorptive state during 3 hours and change after feeding on study day 1
  The examinee is required to say as many words as they can think of in one minute that begin with a given letter of the alphabet. The task contains three trials. Measures phonetic verbal fluency. The raw score (total and mean words recorded across the three trials) was reported.
Group differences in learning and memory as measured by Auditory Verbal Learning Test (AVLT) | Postabsorptive state during 3 hours and change after feeding on study day 1
  a verbal episodic memory test that evaluates a wide diversity of functions: short-term auditory-verbal memory, rate of learning, retention and recognition of information.
Group differences in attention and executive functions as measured by PASAT | Postabsorptive state during 3 hours and change after feeding on study day 1
  a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability.
Group differences in attention and executive functions as measured by Trail Making Test (TMT) | Postabsorptive state during 3 hours and change after feeding on study day 1
  n Part A, the examinee is instructed to connect a set of 25 circles with numbers as quickly as possible while maintaining accuracy. In Part B, the examinee is instructed to connect a set of 25 circles, alternating between numbers and letters, as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and mental flexibility. The total time in seconds was reported for each measure.
Group differences in overall cognitive abilities as measured by Montreal Cognitive Assessment (MoCA) | Postabsorptive state during 3 hours and change after feeding on study day 1
  assesses several cognitive domains and is used for the screening of mild cognitive impairment. Total scores range from 0-30 with lower scores indicating decreased functioning.
Group differences in attention and executive functions as measured by Brief-A | Postabsorptive state during 3 hours and change after feeding on study day 1
  a standardized self-report that captures views of an adult's executive functions or self-regulation in his or her everyday environment.
diet recall | on study day 1
  The subject is asked to recall in detail all the food and drink consumed during the 24 hours prior to the test day.

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, Principal Investigator — Study Principal Investigator
Locations (1):
- Texas A&M University-CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berger MM, Singer P, Wierzchowska-McNew RA, Viana MV, Ben-David IA, Pantet O, Perez C, Thaden JJ, Engelen MPKJ, Deutz NEP. Cytokine response to critical illness and its relation to amino acid metabolism. Clin Nutr. 2025 Sep;52:195-202. doi: 10.1016/j.clnu.2025.07.018. Epub 2025 Jul 26. PMID 40784156
- [Derived] Deutz LN, Wierzchowska-McNew RA, Deutz NE, Engelen MP. Reduced plasma glycine concentration in healthy and chronically diseased older adults: a marker of visceral adiposity? Am J Clin Nutr. 2024 Jun;119(6):1455-1464. doi: 10.1016/j.ajcnut.2024.04.008. Epub 2024 Apr 12. PMID 38616018
- [Derived] Engelen MPKJ, Kirschner SK, Coyle KS, Argyelan D, Neal G, Dasarathy S, Deutz NEP. Sex related differences in muscle health and metabolism in chronic obstructive pulmonary disease. Clin Nutr. 2023 Sep;42(9):1737-1746. doi: 10.1016/j.clnu.2023.06.031. Epub 2023 Jul 26. PMID 37542951
- [Derived] Deutz NEP, Singer P, Wierzchowska-McNew RA, Viana MV, Ben-David IA, Pantet O, Thaden JJ, Ten Have GAM, Engelen MPKJ, Berger MM. Females have a different metabolic response to critical illness, measured by comprehensive amino acid flux analysis. Metabolism. 2023 May;142:155400. doi: 10.1016/j.metabol.2023.155400. Epub 2023 Jan 27. PMID 36717057
- [Derived] Wierzchowska-McNew RA, Engelen MPKJ, Thaden JJ, Ten Have GAM, Deutz NEP. Obesity- and sex-related metabolism of arginine and nitric oxide in adults. Am J Clin Nutr. 2022 Dec 19;116(6):1610-1620. doi: 10.1093/ajcn/nqac277. PMID 36166849
- [Derived] Pinson MR, Deutz NEP, Harrykissoon R, Zachria AJ, Engelen MPKJ. Disturbances in branched-chain amino acid profile and poor daily functioning in mildly depressed chronic obstructive pulmonary disease patients. BMC Pulm Med. 2021 Nov 7;21(1):351. doi: 10.1186/s12890-021-01719-9. PMID 34743729
- [Derived] Deutz NEP, Singer P, Wierzchowska-McNew RA, Viana MV, Ben-David IA, Pantet O, Thaden JJ, Ten Have GAM, Engelen MPKJ, Berger MM. Comprehensive metabolic amino acid flux analysis in critically ill patients. Clin Nutr. 2021 May;40(5):2876-2897. doi: 10.1016/j.clnu.2021.03.015. Epub 2021 Mar 18. PMID 33946038